CLINICAL TRIAL: NCT01214044
Title: Determination of the Circadian Resetting Effects of Escitalopram and Testing for Correlations Between Circadian Resetting and Antidepressant Effects
Brief Title: Circadian Effects of Escitalopram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Jonathan Emens, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LXP-MD-132
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drug (Experimental): Subjects will have a total of 12 visits to Oregon Clinical & Translational Research Institute at Oregon Health & Science University over the 14-16 weeks of study. Subjects will first undergo an initial screening visit to determine eligibility. Subjects who meet criteria and agree to participate will then stop taking their current antidepressant medication (if applicable), during which time the study doctor and staff will conduct weekly mood assessments to ensure safety. Subjects will then have a study initiation/materials visit followed by 9 visits during treatment with placebo or escitalopram. A final post-study follow-up safety visit will be scheduled at the end of treatment.
  Interventions: Drug: placebo/escitalopram

INTERVENTIONS:
Drug: placebo/escitalopram — Subjects will first complete a one week, single-blind placebo lead in phase. Subjects will then receive escitalopram for 8 weeks. Subjects will receive 10 mg/day for the first 2 weeks of active treatment, and then 20 mg/day for the remaining 6 weeks of treatment. Medication will be dispensed on a weekly basis.
  Other Names: Lexapro; escitalopram

SUMMARY:
The goal of the study is to obtain preliminary data that will test whether the antidepressant medication escitalopram resets the body clock: a collection of nerve cells in the brain that control the timing of many body processes. The study will also test whether the improvement in depression symptoms with escitalopram correlates with the degree to which the timing of the body clock is properly aligned with the timing of sleep.

DETAILED DESCRIPTION:
Background: The human biological clock (circadian pacemaker) has long been thought to play a role in non-seasonal depression. A connection is suggested by the demonstration of 24-hour rhythms in mood, subjective and objective changes in sleep with depression, and reports of changes in the timing and amplitude of biological rhythms in depression. Furthermore, it is known that the neurotransmitter serotonin has a significant role in regulating biological rhythms and that drugs that act on serotonin (such as some antidepressants) are able to reset the biological clock in animals.

Objective: The aim of the study is to obtain preliminary data that will test whether the antidepressant medication escitalopram has a resetting effect on the human biological clock and whether the improvement in depression symptoms with escitalopram correlates with the degree to which the timing of the biological clock is realigned with the timing of sleep.

Design: 14-16-week, fixed dose (after titration), open label trial.

Setting and Subjects: 50 individuals will be screened for participation. 15 individuals with unipolar, non-seasonal depression will be studied over 1 year.

Intervention: Subjects will first complete a one week, single-blind placebo lead-in phase. Subjects will then receive escitalopram for 8 weeks (10 mg/day for the first 2 weeks of treatment and then 20mg/day for the remaining 6 weeks of treatment).

Measurements: Subjects will keep a sleep diary and wear a wrist activity monitor throughout the study to document the timing and quality of sleep. On two occasions (end of placebo week and end of last treatment week) blood and/or saliva will be sampled every 30 minutes for 7 hours and the resulting samples will be assayed for melatonin. The onset of melatonin secretion (dim light melatonin onset or DLMO) will be used to mark the timing of the biological clock (circadian phase). Circadian misalignment will be measured using the time interval between the DLMO and the average midsleep of the prior week (phase angle difference or PAD). Mood will be assessed throughout the study using the Hamilton Depression Rating Scale (HAM-D) as well as the Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* able to comply with requirements of the experimental protocol
* competent to sign informed consent
* have mild to severe major depressive disorder without psychotic features and without a seasonal pattern
* currently be under the care of a licensed mental health care provider or primary care physician
* Score > 7 when interviewed by a trained rater using the 21-Item Hamilton Depression Scale (HAM-D)
* be in good physical health
* not be suicidal
* not be taking any other antidepressant medications besides escitalopram during the study
* be free of antidepressant medications for 2-4 weeks prior to beginning the study
* not have a history of transmeridian travel or shift work in the past 2 months and have no plans for transmeridian travel or shift work for the duration of the study
* be able to maintain a regular sleep wake schedule for the weeks one and nine of study
* women of childbearing potential must have a negative pregnancy test and practice an acceptable method of birth control

Exclusion Criteria:

* abnormal heart, liver, or kidney function
* significant laboratory abnormalities on Complete Blood Count, Complete Metabolic Set, Thyroid Stimulating Hormone, EKG, & urinalysis
* shift work or transmeridian travel in the last 2 months
* current use of melatonin
* evidence of a primary sleep disorder by history
* women who are pregnant or lactating
* be taking medications with known sedative or stimulating effects or that would interfere with the production of melatonin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Emens, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug: Subjects will have a total of 12 visits to Oregon Clinical & Translational Research Institute at Oregon Health & Science University over the 14-16 weeks of study. Subjects will first undergo an initial screening visit to determine eligibility. Subjects who meet criteria will then stop taking their current antidepressant medication (if applicable), during which time the study doctor and staff will conduct weekly mood assessments to ensure safety. Subjects will then have a study initiation/materials visit followed by 9 visits during treatment with placebo or escitalopram. A final post-study follow-up safety visit will be scheduled at the end of treatment.
  placebo/escitalopram: Subjects will first complete a one week, single-blind placebo lead in phase. Subjects will then receive escitalopram for 8 weeks. Subjects will receive 10 mg/day for the first 2 weeks of active treatment, and then 20 mg/day for the remaining 6 weeks of treatment. Medication will be dispensed on a weekly basis.
Period: Visit 1: Screening and Consent, Washout
Arm/Group | Study Drug
Started | 31
Completed | 19
Not Completed | 12
Not completed — Withdrawal by Subject | 5
Not completed — Ineligible | 3
Not completed — Lost to Follow-up | 4
Period: Visit 2: End Washout & Start Placebo
Arm/Group | Study Drug
Started | 19
Completed | 17 (2 subjects dropped out during the placebo week (between study visits 2 & 3))
Not Completed | 2
Period: Visits 3-5: Escitalopram 10 mg Daily
Arm/Group | Study Drug
Started | 17
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Visits 6-11: Escitalopram 20 mg Daily
Arm/Group | Study Drug
Started | 14
Completed | 10
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Drug: Subjects will have a total of 12 visits to Oregon Clinical & Translational Research Institute at Oregon Health & Science University over the 14-16 weeks of study. An initial screening visit will determine eligibility. Subjects who meet criteria and agree to participate will then stop taking their current antidepressant medication (if applicable), during which time the study doctor and staff will conduct weekly mood assessments to ensure safety. Subjects will then have a study initiation/materials visit followed by 9 visits during treatment with placebo or escitalopram. A final post-study follow-up safety visit will be scheduled at the end of treatment.
  Placebo/escitalopram: Subjects will first complete a one week, single-blind placebo lead in phase. Subjects will then receive escitalopram for 8 weeks. Subjects will receive 10 mg/day for the first 2 weeks of active treatment, and then 20 mg/day for the remaining 6 weeks of treatment. Medication will be dispensed weekly.
Arm/Group | Study Drug
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Dim Light Melatonin Onset
Description: The Dim Light Melatonin Onset (DLMO) is the time of the onset of melatonin secretion under dim light conditions using the equivalent thresholds of 10 pg/ml in plasma and 3 pg/ml in saliva. It is a marker of biological time. Data are provided in decimal and military time (e.g., 9:30 pm equals 21.50).
  This measure is used to determine if there was a change in the time of the dim light melatonin onset (DLMO) before treatment with escitalopram (at Study Visit 3) and after treatment with escitalopram (at Study Visit 11).
Time Frame: 8 Weeks: Study Visit 3 (after 1 week of placebo) to study Visit 11 (after 8 weeks of escitalopram)
Population: Of the 10 subjects who completed all study procedures, adequate dim light melatonin data from both study visits 3 and 11 were available for 9 subjects.
Measure: Mean (Standard Deviation); unit: decimal military time (hours)
Arm/Group | Study Drug
Number analyzed (Participants) | 9
decimal military time (hours)
  Baseline DLMO | 21.17 (1.24)
  Post-escitalopram DLMO | 20.77 (1.17)
Statistical Analysis 1: Comparison: Study Drug; A within subjects comparison was done to compare the time of the dim light melatonin onset before treatment with escitalopram (Study Visit 3) and after treatment with escitalopram (Study Visit 11); Test type: Other — A paired t-test was done to see if the time of the dim light melatonin onset changed from baseline to post-treatment; p = 0.2, t-test, 2 sided — A priori threshold for significance was p = 0.05; paired t-test

2. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Scores
Description: The HAM-D is the total score on the 21-question Hamilton Depression Rating Scale. Scores range from 0 to 53 with higher scores indicating worse symptoms of depression.
Time Frame: 8 Weeks: Study Visit 3 (after 1 week of placebo) to study Visit 11 (after 8 weeks of escitalopram)
Population: Of the 10 subjects who completed all study procedures, adequate Hamilton Depression Rating Scale data from both study visits 3 and 11 were available for 7 subjects.
Measure: Mean (Standard Deviation); unit: units on scale (scores)
Groups:
- Study Drug: Subjects will have a total of 12 visits to Oregon Clinical & Translational Research Institute at Oregon Health & Science University over the 14-16 weeks of study. An initial screening visit will determine eligibility. Subjects who meet criteria and agree to participate will then stop taking their current antidepressant medication (if applicable), during which time the study doctor and staff will conduct weekly mood assessments to ensure safety. Subjects will then have a study initiation/materials visit followed by 9 visits during treatment with placebo or escitalopram. A final post-study follow-up safety visit will be scheduled at the end of treatment.
  placebo/escitalopram: Subjects will first complete a one week, single-blind placebo lead in phase. Subjects will then receive escitalopram for 8 weeks. Subjects will receive 10 mg/day for the first 2 weeks of active treatment, and then 20 mg/day for the remaining 6 weeks of treatment. Medication will be dispensed on a weekly basis.
Arm/Group | Study Drug
Number analyzed (Participants) | 7
units on scale (scores) | -2.3 (2.0)
Statistical Analysis 1: Comparison: Study Drug; We hypothesized that there would be a decrease in the Hamilton-21 score with escitalopram treatment. A within subjects comparison was done to compare the Hamilton-21 score before treatment with escitalopram (Study Visit 3) and after treatment with escitalopram (Study Visit 11); Test type: Other — A paired t-test was done to see if the Hamilton-21 score decreased from baseline to post-treatment; p = 0.01, t-test, 1 sided — A priori threshold for significance was p = 0.05; paired t-test

3. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II) Scores
Description: The BDI-II is the total score on the 21-question Beck Depression Inventory II questionnaire. Scores range from 0 to 63 with higher scores indicating worse symptoms of depression.
Time Frame: 8 Weeks: Study Visit 3 (after 1 week of placebo) to study Visit 11 (after 8 weeks of escitalopram)
Population: Of the 10 subjects who completed all study procedures, Beck Depression Inventory-II data from both study visits 3 and 11 were available for 7 subjects.
Measure: Mean (Standard Deviation); unit: units on scale (scores)
Arm/Group | Study Drug
Number analyzed (Participants) | 7
units on scale (scores) | -3.3 (7.4)
Statistical Analysis 1: Comparison: Study Drug; We hypothesized that there would be a decrease in the Beck Depression Inventory-II score with escitalopram treatment. A within subjects comparison was done to compare the Beck Depression Inventory-II score before treatment with escitalopram (Study Visit 3) and after treatment with escitalopram (Study Visit 11); Test type: Other — A paired t-test was done to see if the Beck Depression Inventory-II score decreased from baseline to post-treatment; p = 0.14, t-test, 1 sided — A priori threshold for significance was p = 0.05; paired t-test

4. Secondary Outcome: Change in Phase Angle Difference (PAD)
Description: The PAD is the time interval (number of hours) between the Dim Light Melatonin Onset (DLMO) and the average midpoint of sleep during the prior week. Larger PADs indicate a longer time interval between the DLMO and midpoint of sleep. A negative change in PAD value indicates a shortening of the time interval from Study Visit 3 to Study Visit 11.
Time Frame: 8 Weeks: Study Visit 3 (after 1 week of placebo) to study Visit 11 (after 8 weeks of escitalopram)
Population: Of the 10 subjects who completed all study procedures, adequate PAD data from both study visits 3 and 11 (derived from dim light melatonin onset and sleep diary) were available for 7 subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Study Drug
Number analyzed (Participants) | 7
hours | -0.6 (0.8)
Statistical Analysis 1: Comparison: Study Drug; We hypothesized that there would be a correlation between the change in phase angle difference and the decrease in the Hamilton-21 score with escitalopram treatment. The phase angle difference is the interval, in hours, between the dim light melatonin onset (a marker of biological time) and the average midpoint of sleep during the prior week; Test type: Other — Spearman's rank-order correlation (non-parametric test) was used; p = 0.06, Spearman's rank-order correlation — Spearman's rho (rs) = 0.66
Statistical Analysis 2: Comparison: Study Drug; We hypothesized that there would be a correlation between the change in phase angle difference and the decrease in the Beck Depression Inventory-II score with escitalopram treatment. The phase angle difference is the interval, in hours, between the dim light melatonin onset (a marker of biological time) and the average midpoint of sleep during the prior week; Test type: Other — Spearman's rank-order correlation (non-parametric test) was used; p = 0.48, Spearman's rank-order correlation — Spearman's rho (rs) = 0.02

ADVERSE EVENTS:
Time Frame: Participants were assessed over 14 weeks (or 16 weeks in two subjects who were on fluoxetine at enrollment and therefore had a 4-week, instead of a 2-week, washout period per the protocol). Subjects had a weekly contact with study personnel throughout the 14 or 16 weeks of study except for the two week medication taper period between the last two study visits.
Groups:
- Visit 1: Screening & Consent, Washout: Subjects will have a total of 12 visits to Oregon Clinical & Translational Research Institute at Oregon Health & Science University over the 14-16 weeks of study. An initial screening visit will determine eligibility. Subjects who meet criteria and agree to participate will then stop taking their current antidepressant medication (if applicable), during which time the study doctor and staff will conduct weekly mood assessments to ensure safety.
- Visit 2: End Washout & Start Placebo: After completing the washout period, Subjects will then complete a one week, single-blind placebo lead in phase.
- Visits 3-5: Escitalopram 10 mg Daily: After the week of placebo, Subjects will then receive 10 mg/day of escitalpram for the first 2 weeks of active treatment.
- Visits 6-11: Escitalopram 20 mg Daily: After receiving 10 mg/day of escitalopram for 2 weeks, subjects will then receive escitalopram, 20 mg/day for the remaining 6 weeks of treatment.
Arm/Group | Visit 1: Screening & Consent, Washout | Visit 2: End Washout & Start Placebo | Visits 3-5: Escitalopram 10 mg Daily | Visits 6-11: Escitalopram 20 mg Daily
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/19 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/19 | 0/17 | 1/14
Other Adverse Events (participants affected / at risk) | 0/31 | 0/19 | 1/17 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visit 1: Screening & Consent, Washout (N=31) | Visit 2: End Washout & Start Placebo (N=19) | Visits 3-5: Escitalopram 10 mg Daily (N=17) | Visits 6-11: Escitalopram 20 mg Daily (N=14)
suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — In this cohort of subjects with mild to severe Major Depressive Disorder, one subject was admitted to an outside hospital following a suicide attempt and was subsequently transferred to outpatient facility for ongoing treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visit 1: Screening & Consent, Washout (N=31) | Visit 2: End Washout & Start Placebo (N=19) | Visits 3-5: Escitalopram 10 mg Daily (N=17) | Visits 6-11: Escitalopram 20 mg Daily (N=14)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One subject reported the onset of a headache around 6 pm with subsequent feelings of her heart racing, feeling flushed in her face & neck and some itchiness. The symptoms resolved after 2 hours.

LIMITATIONS AND CAVEATS:
The sample size was small because this was a preliminary study that aimed to collect pilot data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-09-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT01214044/Prot_SAP_000.pdf